CLINICAL TRIAL: NCT06956092
Title: Prospective Clinical Study of Glofitamab for Consolidation After First-line Treatment of High-risk Large B-cell Lymphoma
Brief Title: Glofitamab for Consolidation After First-line Treatment of High-risk Large B-cell Lymphoma
Acronym: Glofitamab
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Professor, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-IIT-0013
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: B Cell Lymphoma (BCL)
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Glofitamab treatment (Experimental)
  Interventions: Biological: Glofitamab treatment

INTERVENTIONS:
Biological: Glofitamab treatment — eceive Glofitamab treatment as per the instructions in the package insert.

SUMMARY:
The goal of this clinical trial is to learn if Glofitamab works for consolidation after first-line treatment of high-risk Large B-cell Lymphoma (LBCL). It will also learn about the safety of Glofitamab treatment. The main questions it aims to answer are:

* Does Glofitamab treatment result in prolonged clinical benefit to patients with high-risk LBCL after first-line treatment?
* What medical problems do participants have when receiving Glofitamab treatment?

In this investigator-initiated, single-arm clinical trial, participants will:

* Receive Glofitamab treatment as per the instructions in the package insert.
* Visit the clinic as instructed for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form.
2. Age 18-75 years (inclusive, including 18 and 75 years) at screening; no restriction on gender.
3. Diagnosed with B-cell non-Hodgkin lymphoma according to the 2022 WHO Classification of Tumors of Hematopoietic and Lymphoid Tissues (5th edition). The following subtypes are included in this trial:

1) Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS), defined as high-risk disease meeting at least one of the following criteria: IPI score of 4-5 at initial diagnosis, TP53 negativity or overexpression (>50%) or TP53 mutation identified by gene sequencing, MYC rearrangement, CD5(+), MYC and BCL2 co-expression.

2) Follicular lymphoma-transformed large B-cell lymphoma. 3) High-grade B-cell lymphoma (HGBL) with MYC and BCL2 rearrangement. 4) High-grade B-cell lymphoma, not otherwise specified (HGBL-NOS). 5) Intravascular large B-cell lymphoma. 6) Large tumor mass (≥7.5 cm). 4. Histopathologically and/or cytologically confirmed CD20-positive large B-cell lymphoma patients who have achieved CR, Cru, or VGPR after prior first-line treatment with rituximab-containing chemoimmunotherapy.

5. Expected survival ≥12 weeks. 6. Target lesion defined as a lymph node-based lesion with a long diameter ≥15 mm or an extranodal lesion >10 mm (according to Lugano 2014 criteria); lesions previously treated with radiotherapy must show clear progression post-radiation to be considered measurable.

7. Patients with occult or early-stage hepatitis B infection (defined as HBcAb positive and HBsAg negative) are eligible for inclusion if HBV DNA PCR testing is negative. These patients will undergo monthly HBV DNA PCR monitoring. Patients seropositive for HCV antibodies are eligible if HCV RNA PCR testing is negative.

8. Adequate bone marrow reserve, defined as: neutrophil count ≥1.0×10^9/L; lymphocyte count ≥0.2×10^9/L; hemoglobin >80 g/L; platelets >80×10^9/L.

9. Non-hematologic toxicities caused by prior treatments (excluding disease-related conditions) must have resolved to ≤Grade 1 prior to enrollment (except alopecia and chemotherapy-induced Grade ≥2 neurotoxicity).

10. Appropriate organ function, meeting the following criteria (excluding abnormalities caused by tumor infiltration):

* Aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN); alanine aminotransferase (ALT) ≤3 times ULN; total serum bilirubin ≤2 times ULN, unless Gilbert syndrome is present. Patients with Gilbert syndrome can be included if total bilirubin ≤3 times ULN and direct bilirubin ≤1.5 times ULN.
* Serum creatinine ≤1.5 times ULN or creatinine clearance ≥60 mL/min (using Cockcroft-Gault formula: Male CrCl = [(140-age) × weight (kg)] / [0.818 × creatinine (μmol/L)]; Female CrCl = [(140-age) × weight (kg) × 0.85] / [0.818 × creatinine (μmol/L)]).
* Minimum pulmonary reserve: ≤Grade 1 dyspnea (CTCAE v5.0) and oxygen saturation ≥92% under non-oxygenated conditions.
* Left ventricular ejection fraction (LVEF) ≥50% by echocardiography; no clinically significant ECG abnormalities; no clinically significant pericardial effusion or pleural effusion.
* International normalized ratio (INR) ≤1.5 times ULN and activated partial thromboplastin time (APTT) ≤1.5 times ULN.

  11. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 12. No central nervous system lymphoma determined by cranial MRI. 13. Women of childbearing potential must have a negative blood/urine pregnancy test within 7 days prior to infusion. All male and female patients capable of reproduction must agree to use effective contraception throughout the study and for at least 2 years after study treatment administration. A patient is deemed capable of reproduction based on their biological ability to conceive and normal sexual activity, as judged by the investigator. Women are deemed incapable of reproduction if they meet at least one of the following criteria: medically-confirmed ovarian failure, hysterectomy, bilateral oophorectomy, or post-menopausal status (defined as cessation of menstruation for at least 12 consecutive months).

Exclusion Criteria:

**Exclusion Criteria:**

1. History of severe allergy or hypersensitivity reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins).
2. Received autologous hematopoietic stem cell transplantation (ASCT) within 100 days prior to the first dose of Glofitamab; received chimeric antigen receptor T-cell (CAR-T) therapy within 30 days prior to the first dose of Glofitamab.
3. Previously underwent allogeneic stem cell transplantation or allogeneic CAR-T therapy.
4. History of solid organ transplantation.
5. History of acute or chronic active hepatitis B or hepatitis C infection. Patients with a history of hepatitis must demonstrate viral clearance based on standard serological and genetic testing (i.e., hepatitis B surface antibody positive, other markers negative, and HBV DNA PCR negative) to be eligible; other cases require approval from the medical monitor.
6. Infection with human immunodeficiency virus (HIV).
7. Known or suspected chronic active Epstein-Barr virus (CAEBV) infection.
8. Presence of uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding nail bed fungal infections) at screening or occurrence of any serious infection within 4 weeks prior to the first infusion of Glofitamab (as judged by the investigator).
9. Current or history of central nervous system (CNS) disorders such as seizures, ischemic/hemorrhagic cerebrovascular events, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychiatric disorders, or autoimmune diseases involving the CNS.
10. History of autoimmune diseases, including but not limited to: myasthenia gravis, polymyositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-associated vascular thrombosis, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, glomerulonephritis, or active autoimmune cytopenias (autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]).

    * Patients with long-standing or well-controlled autoimmune diseases may be eligible after discussion and confirmation with the investigator.
    * Patients with autoimmune thyroid dysfunction receiving stable doses of thyroid replacement hormone may be eligible.
    * Patients with well-controlled Type 1 diabetes (defined as fasting HbA1c <8% at screening and no ketoacidosis) are eligible.
    * Patients with skin-limited conditions such as eczema, psoriasis, chronic lichen simplex, or vitiligo may be eligible if the following criteria are met:

      * Rash involves <10% of body surface area.
      * Disease is well-controlled at baseline and requires only low-dose topical corticosteroids.
      * No exacerbations requiring treatment with psoralen plus UVA light, methotrexate, retinoids, biologics, oral calcineurin inhibitors, high-dose or systemic corticosteroids during the past 12 months.
11. Presence of primary or secondary active CNS lymphoma (patients with symptoms suggestive of CNS involvement must undergo lumbar puncture and MRI to exclude CNS lymphoma).
12. Prior receipt of other genetically modified T-cell therapy or CAR-T therapy.
13. Diagnosis of progressive multifocal leukoencephalopathy (PML).
14. Clinical emergencies requiring urgent intervention due to lymphoma-related obstruction or compression, such as intestinal obstruction or vascular compression, at screening.
15. Cardiac conditions meeting any of the following: left ventricular ejection fraction (LVEF) ≤45% (by echocardiography); New York Heart Association (NYHA) class III or IV congestive heart failure; severe arrhythmias requiring treatment, including QTc interval ≥450ms for males or ≥470ms for females (QTcB=QT/RR^1/2); uncontrolled hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg), pulmonary hypertension, or unstable angina; history of cardiac angioplasty or stent placement, myocardial infarction, unstable angina, or other clinically significant cardiac conditions within 12 months prior to administration; clinically significant valvular disease; lymphoma involving atrial or ventricular structures; or other cardiac diseases deemed unsuitable by the investigator.
16. Thromboembolic events (such as deep vein thrombosis or pulmonary embolism) within 6 months prior to screening.
17. Malignancies other than those indicated for this trial within 5 years prior to screening, except for melanoma, skin carcinoma, or in-situ cancers (e.g., cervical, bladder, breast carcinoma).
18. Receipt of live attenuated vaccines within 4 weeks prior to the first infusion of Glofitamab or expected need for such vaccines during the study period.
19. Major surgery within 4 weeks prior to the first infusion of Glofitamab. Protocol-required procedures such as tumor biopsy and bone marrow biopsy are allowed.
20. Systemic immunosuppressive therapy (including but not limited to azathioprine, methotrexate, thalidomide, or anti-TNF agents) within 2 weeks prior to the first infusion of Glofitamab. Corticosteroid therapy at ≤25 mg/day prednisone or equivalent is permitted.

    * Inhaled and topical corticosteroids are allowed.
21. Inability to comply with protocol-mandated hospitalization and activity restrictions.
22. Pregnant or breastfeeding women, or male or female patients of childbearing potential who refuse to use effective contraception during the study and for 2 years after the cellular infusion.
23. Participation in another interventional clinical trial, receipt of investigational drugs, or intent to enroll in another trial or receive non-protocol-defined antitumor therapy within 3 months before Glofitamab administration.
24. Any severe medical condition or laboratory abnormality, as determined by the investigator or medical monitor, that could compromise patient safety, adherence to the protocol, or interpretation of results.
25. Investigator deems the patient unsuitable for this trial (e.g., poor compliance, substance abuse, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
two year PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Department of Oncology, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No